CLINICAL TRIAL: NCT02994667
Title: Pacemaker Utilization and Ventricular Pacing in Patients Undergoing Trans-catheter Aortic Valve Replacement (TAVR)
Acronym: PPM in TAVR
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 014-286
Record Dates: First submitted 2016-11-18; First posted 2016-12-16 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Ventricular Flutter; Atrioventricular Block; Intraventricular Conduction Delay; Bundle Branch Block; Pacemaker Implantation
Keywords: Electrophysiology
MeSH Terms: conditions — Ventricular Flutter; Atrioventricular Block; Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker After TAVR: The study cohort will comprise all consecutive patients who undergo permanent pacemaker placement for new conduction disturbances after TAVR at THHBP between 1/1/2015 and 12/31/2016.
  Interventions: Device: Permanent Pacemaker Placement

INTERVENTIONS:
Device: Permanent Pacemaker Placement

SUMMARY:
The purpose of this study is to assess the incidence (at 90-days) of ventricular pacing in patients undergoing permanent pacemaker placement after TAVR.

As well as incidence (at 90-days) of atrioventricular block (AVB), intraventricular conduction delay (IVCD), bundle branch block (BBB), and rate histogram in patients undergoing permanent pacemaker placement after TAVR.

DETAILED DESCRIPTION:
Development of atrioventricular (AV) conduction system abnormalities requiring placement of a permanent pacemaker (PPM) is a known complication of transcatheter aortic valve replacement (TAVR). Male gender, pre-existing AV conduction system abnormalities, transient AV block intra-procedurally, and use of a self-expanding valve have all been associated with increased risk of AV block and need for permanent pacemaker placement. Persistent AV conduction abnormalities have been documented in approximately 15% of patients who receive an Edwards Sapien valve, with 4% requiring permanent pacemaker placement. 22-28% of patients who receive a CoreValve require permanent pacemaker placement in some studies. In one study, 78% of patients who underwent His bundle electrogram assessment during CoreValve placement had transient or persistent AV conduction system abnormalities during the procedure.

Pacemakers placed at The Heart Hospital Baylor Plano are produced by two manufactures: Medtronic, Inc. and St. Jude Medical, Inc. Each of these manufacturers have pacemakers with algorithms designed to minimize right ventricular pacing. Medtronic's algorithm is referred to as "MVP" (Managed Ventricular Pacing), and St. Jude Medical's algorithm is referred to as "VIP" (Ventricular Intrinsic Preference). Each of these techniques purports to reduce unnecessary right ventricular (RV) pacing through a novel pacemaker algorithm. Both manufacturers' pacemaker programmers and remote monitoring systems allow for demonstration of the percentage of ventricular pacing performed by the device.

The Investigators propose to assess the 90 day- ventricular pacing, atrioventricular block (AVB), intraventricular conduction delay (IVCD), bundle branch block (BBB), and rate histogram incidence in those patients who undergo pacemaker implantation due to elevated risk (or occurrence of) high-grade AV block after TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients undergoing Transcatheter Aortic Valve Replacement
* Indication for PPM including:

  1. Persistent 3rd degree AVB
  2. Transient 3rd degree AVB
  3. New Left BBB
  4. New bifascicular block
  5. New first degree AV block
  6. Any conduction disturbance determined by the investigator to be related to the TAVR procedure 4. Patients receiving post-TAVR PPM with one of the following devices

  a. Medtronic: i. ADAPTA DR -ADDR01 ii. ADAPTA L DR-ADDRL1 iii. ADVISA MRI-A2DR01 b. St. Jude Medical: i. Zypher 5820 ii. Zypher 5826 iii. Accent pm2110 iv. Accent pm2210 v. Assurity pm2240 vi. Endurity Pm2160

Exclusion Criteria:

* Pregnancy-Women of childbearing potential should have negative urine 'pregnancy test prior to enrollment
* Patients with implanted pacemaker
* Patients with implantable cardiac defibrillator
* Indication for post TAVR PPM not related to the procedure including sinus node dysfunction/sick sinus syndrome.
* Medically unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will comprise all consecutive patients who undergo permanent pacemaker placement for new conduction disturbances after TAVR at THHBP between 1/1/2015 and 12/31/2016 and will consist of up to 50 patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Ventricular Pacing | 7-90 days
  Incidence of Ventricular pacing post permanent pacemaker placement after TAVR as indicated by Pacemaker interrogation or remote monitoring system.

SECONDARY OUTCOMES:
Incidence of other conduction disturbances | 7-90 days
  Freedom from documented atrioventricular block (AVB), intraventricular conduction dely (IVCD), bundle branch block (BBB) as indicated by pacemaker interrogation or remote monitoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Deville, MD, Principal Investigator — The Heart Hospital Baylor of Plano
Locations (1):
- The Heart Hospital Baylor of Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data on the clinical and non-clinical risk factors will be summarized using means, standard deviations (SDs) and percentages. The Kaplan-Meier method will be used to construct a ventricular pacing free curve summarizing time-to ventricular pacing incidence in the study cohort -the competing risk of death will be accounted in the analysis.